CLINICAL TRIAL: NCT03953196
Title: A Phase 0 Study Exploring the Use of Vaccine and Antigen Challenges for Immune Monitoring in Healthy Volunteers
Brief Title: A Study Exploring the Use of Vaccine and Antigen Challenges for Immune Monitoring in Healthy Participants
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CR108590; NOPRODNAP0016 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-04-01; First posted 2019-05-16 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic; Endotoxins; Yeast, Dried

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Cohort 1: Vaccine Challenge Imvanex (Experimental): Participants will receive single dose of Imvanex subcutaneously on Day 1. Participants will also be included in the DREEM EEG substudy.
  Interventions: Biological: Imvanex
- Cohort 2: Vaccine Challenge Shingrix (Experimental): Participants will receive single dose of Shingrix intramuscularly on Day 1. Participants will also be included in the DREEM EEG substudy.
  Interventions: Biological: Shingrix
- Cohort 3: Antigen Challenge Lipopolysaccharides (LPS) (Experimental): Participants will receive a single dose of LPS intravenously (IV) on Day 1. Participants will also be included in the DREEM EEG substudy and vital patch physIQ platform substudy.
  Interventions: Biological: LPS
- Cohort 4: Antigen Challenge Candin (Experimental): Participants will receive one single injection of Candin and one single injection of saline control intradermally on Day 1. Participants will also be included in the DREEM EEG substudy.
  Interventions: Biological: Candin; Other: Saline Control
- Cohort 5: Skin Wounding Challenge (Experimental): 3 punch biopsies will be performed per standard dermatologic practice guidelines. Lower abdomen tissue biopsy specimens will be collected on Day 1.
  Interventions: Other: Skin Biopsy

INTERVENTIONS:
Biological: Imvanex — Imvanex 0.5 milliliter (mL) suspension for injection will be administered as single subcutaneous (SC) injection.
  Other Names: Imvamune
  Arms: Cohort 1: Vaccine Challenge Imvanex
Biological: Shingrix — Shingrix 0.5 mL suspension will be administered as single intramuscular (IM) injection.
  Arms: Cohort 2: Vaccine Challenge Shingrix
Biological: LPS — LPS 1.0 nanogram per kilogram (ng/kg) endotoxin suspension will be administered as single IV injection.
  Other Names: Endotoxin
  Arms: Cohort 3: Antigen Challenge Lipopolysaccharides (LPS)
Biological: Candin — Candin 0.1 mL solution for injection will be administered as one intradermal injection.
  Other Names: Candida albicans
  Arms: Cohort 4: Antigen Challenge Candin
Other: Skin Biopsy — 3 punch biopsies will be performed and lower abdomen tissue biopsy specimens will be collected on Day 1.
  Arms: Cohort 5: Skin Wounding Challenge
Other: Saline Control — Saline control solution for injection will be administered as one intradermal injection.
  Arms: Cohort 4: Antigen Challenge Candin

SUMMARY:
The purpose of this study is to characterize the immune response in vivo using approved vaccines and antigen challenges, as well as a skin wounding challenge to stimulate the immune system.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) between 18 and 30 kilogram per square meter (kg/m^2) (BMI = weight/height^2), inclusive, and a body weight of no less than 50 kilogram (kg)
* Healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) (for Cohort 3) performed at screening. Any abnormalities, must be considered not clinically significant and this determination must be recorded in the participant's source documents and initialed by the investigator
* Healthy on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel, blood coagulation, hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the investigator
* Must sign an informed consent form (ICF) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study
* All women must have a negative highly sensitive serum (Beta-human chorionic gonadotropin [Beta-hCG]) pregnancy test at screening and a negative urine pregnancy test predose on Day 1

Exclusion Criteria:

* History of any type of immunodeficiency or autoimmune disease or disease treatment associated with immune suppression or lymphopenia. These include but are not limited to bone marrow or organ transplantation, lymphoproliferative disorders, T- or B-cell deficiency syndromes, splenectomy, functional asplenia and chronic granulomatous disease
* History of liver or renal insufficiency, significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, bleeding disorders, rheumatologic, psychiatric, or metabolic disturbances, and atopic dermatitis
* Known allergies, hypersensitivity, or intolerance to any of the interventions in this study or their excipients
* History of severe allergic reaction, angioedema, or anaphylaxis to drugs or food
* Contraindications to the use of any of the study interventions per prescribing information

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2019-12-26 (Actual); Study Completion 2019-12-26 (Actual)

PRIMARY OUTCOMES:
Cohort 1 and Cohort 2: Change from Baseline of Immune Cell Populations | Baseline up to 90 days
  Change from baseline in immune cell populations will be measured in peripheral blood samples or tissues of healthy volunteers.
Cohort 3 and Cohort 4: Change from Baseline of Immune Cell Populations | Baseline up to 14 days
  Change from baseline in immune cell populations will be measured in peripheral blood samples or tissues of healthy volunteers.
Cohort 5: Change from Baseline of Immune Cell Populations | Baseline up to 10 days
  Change from baseline in immune cell populations will be measured in tissues of healthy volunteers.
Cohort 1 and Cohort 2: Change from Baseline in Cell Surface Antigen Phenotype | Baseline up to 90 days
  Change from baseline in cell surface antigen phenotype will be measured in peripheral blood samples or tissues of healthy volunteers.
Cohort 3 and Cohort 4: Change from Baseline in Cell Surface Antigen Phenotype | Baseline up to 14 days
  Change from baseline in cell surface antigen phenotype will be measured in peripheral blood samples or tissues of healthy volunteers.
Cohort 5: Change from Baseline in Cell Surface Antigen Phenotype | Baseline up to 10 days
  Change from baseline in cell surface antigen phenotype will be measured in tissues of healthy volunteers.
Cohort 1 and Cohort 2: Change from Baseline in Activation Status of Inflammatory Mediators (Soluble Cytokines and Chemokines) | Baseline up to 90 days
  Soluble cytokines and chemokines will be measured by immunoassay.
Cohort 3 and Cohort 4: Change from Baseline in Activation Status of Inflammatory Mediators (Soluble Cytokines and Chemokines) | Baseline up to 14 days
  Soluble cytokines and chemokines will be measured by immunoassay.
Cohort 5: Change from Baseline in Activation Status of Inflammatory Mediators (Soluble Cytokines and Chemokines) | Baseline up to 10 days
  Soluble cytokines and chemokines will be measured by immunoassay.
Cohort 1 and Cohort 2: Change from Baseline in Activation Status of Inflammatory Mediators (Cell-bound and Tissue-associated Proteins) | Baseline up to 90 days
  Cell-bound and tissue-associated proteins will be measured by established methods including flow cytometry and immunohistochemistry.
Cohort 3 and Cohort 4: Change from Baseline in Activation Status of Inflammatory Mediators (Cell-bound and Tissue-associated Proteins) | Baseline up to 14 days
  Cell-bound and tissue-associated proteins will be measured by established methods including flow cytometry and immunohistochemistry.
Cohort 5: Change from Baseline in Activation Status of Inflammatory Mediators (Cell-bound and Tissue-associated Proteins) | Baseline up to 10 days
  Cell-bound and tissue-associated proteins will be measured by established methods including flow cytometry and immunohistochemistry.
Cohort 1 and Cohort 2: Change from Baseline in Expression of Inflammatory Mediators | Baseline up to 90 days
  Transcriptional changes in gene expression will be measured by established methods such as ribonucleic acid (RNA) microarray, RNAseq, and single cell RNA sequencing, and will be reported in number of gene transcripts per sample or per cell.
Cohort 3 and Cohort 4: Change from Baseline in Expression of Inflammatory Mediators | Baseline up to 14 days
  Transcriptional changes in gene expression will be measured by established methods such as ribonucleic acid (RNA) microarray, RNAseq, and single cell RNA sequencing, and will be reported in number of gene transcripts per sample or per cell.
Cohort 5: Change from Baseline in Expression of Inflammatory Mediators | Baseline up to 10 days
  Transcriptional changes in gene expression will be measured by established methods such as RNA microarray, RNAseq, and single cell RNA sequencing, and will be reported in number of gene transcripts per sample or per cell.

SECONDARY OUTCOMES:
Change in Standard Deviation from Baseline of Immune Cell Populations Within a Participant | Cohort 1 and Cohort 2: Baseline up to 90 days; Cohort 3 and Cohort 4: Baseline up to 14 days; Cohort 5: Baseline up to 10 days
  Change in standard deviation from baseline of immune cell populations within a participant will be measured.
Change in Standard Deviation from Baseline of Immune Cell Populations Between Participants | Cohort 1 and Cohort 2: Baseline up to 90 days; Cohort 3 and Cohort 4: Baseline up to 14 days; Cohort 5: Baseline up to 10 days
  Change in standard deviation from baseline of immune cell populations between participants will be measured.
Change in Standard Deviation from Baseline in Cell Surface Antigen Phenotype Within a Participant | Cohort 1 and Cohort 2: Baseline up to 90 days; Cohort 3 and Cohort 4: Baseline up to 14 days; Cohort 5: Baseline up to 10 days
  Change in standard deviation from baseline in cell surface antigen phenotype within a participant will be measured.
Change in Standard Deviation from Baseline in Cell Surface Antigen Phenotype Between Participants | Cohort 1 and Cohort 2: Baseline up to 90 days; Cohort 3 and Cohort 4: Baseline up to 14 days; Cohort 5: Baseline up to 10 days
  Change in standard deviation from baseline in cell surface antigen phenotype between participants will be measured.
Change in Standard Deviation from Baseline in Activation Status of Inflammatory Mediators Within a Participant | Cohort 1 and Cohort 2: Baseline up to 90 days; Cohort 3 and Cohort 4: Baseline up to 14 days; Cohort 5: Baseline up to 10 days
  Change in standard deviation from baseline in activation status of inflammatory mediators within a participant will be measured.
Change in Standard Deviation from Baseline in Activation Status of Inflammatory Mediators Between Participants | Cohort 1 and Cohort 2: Baseline up to 90 days; Cohort 3 and Cohort 4: Baseline up to 14 days; Cohort 5: Baseline up to 10 days
  Change in standard deviation from baseline in activation status of inflammatory mediators between participants will be measured.
Change in Standard Deviation from Baseline in Expression of Inflammatory Mediators Within a Participant | Cohort 1 and Cohort 2: Baseline up to 90 days; Cohort 3 and Cohort 4: Baseline up to 14 days; Cohort 5: Baseline up to 10 days
  Change in standard deviation from baseline in expression of inflammatory mediators within a participant will be measured.
Change in Standard Deviation from Baseline in Expression of Inflammatory Mediators Between Participants | Cohort 1 and Cohort 2: Baseline up to 90 days; Cohort 3 and Cohort 4: Baseline up to 14 days; Cohort 5: Baseline up to 10 days
  Change in standard deviation from baseline in expression of inflammatory mediators between participants will be measured.
Correlation of Baseline Immune Cell Populations with Vaccine/Antigen Immune Response Phenotype | Cohort 1 and Cohort 2: Baseline up to 90 days; Cohort 3 and Cohort 4: Baseline up to 14 days
  Correlation of baseline immune cell populations with vaccine/antigen immune response phenotype will be measured by phenotypic and functional assays.
Correlation of Genomics with Vaccine/Antigen Immune Response Phenotype | Cohort 1 and Cohort 2: Baseline up to 90 days; Cohort 3 and Cohort 4: Baseline up to 14 days
  Correlation of genomics with vaccine/antigen immune response phenotype will be measured by phenotypic and functional assays.
Correlation of Serology with Vaccine/Antigen Immune Response Phenotype | Cohort 1 and Cohort 2: Baseline up to 90 days; Cohort 3 and Cohort 4: Baseline up to 14 days
  Correlation of serology with vaccine/antigen immune response phenotype will be measured by phenotypic and functional assays.
Correlation of Soluble Proteins with Vaccine/Antigen Immune Response Phenotype | Cohort 1 and Cohort 2: Baseline up to 90 days; Cohort 3 and Cohort 4: Baseline up to 14 days
  Correlation of soluble proteins with vaccine/antigen immune response phenotype will be measured by phenotypic and functional assays.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency